CLINICAL TRIAL: NCT00211471
Title: Treatment of Rubeosis Iridis With Open-Label Anecortave Acetate Sterile Suspension (15mg.).
Brief Title: Treatment of Rubeosis Iridis With Open-Label Anecortave Acetate Sterile Suspension ( 15 mg.).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rubeosis iridis
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Severe Diabetic Retinopathy; Central Retinal Vein Occlusion; Chronic Inflammation; Infectious Diseases
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion; Communicable Diseases | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anecortave acetate

SUMMARY:
To provide use of Anecortave Acetate Sterile Suspension of 15mg for a series of five patients with rubeosis iridis. Rubeosis iridis refers to neovascularization of the iris. It is caused by a number of conditions which include, but are not limited to severe diabetic retinopathy, central retinal vein occlusion, chronic inflammation, and infection. Anecortave acetate is an angiostatic, experimental drug that is being tested to prevent the growth of blood vessels under the retina in patients with age-related macular degeneration (AMD). Therefore, it is logical to apply the usage of Anecortave to patient's with rubeosis iridis in order to reduce the neovascularization stimulus and cause the regression of the abnormal iris vessels.

DETAILED DESCRIPTION:
Patients will receive an injection of 15 mg of Anecortave acetate behind the eye to be treated ("study eye"). They will be evaluated every six months to determine if their condition is stable or worse. Following the injection of study medication, patients will not be required to come in to see the study physician. The investigator or study staff will call the patients on the day following injection to make sure there were no adverse effects to the injection. Patients will then come in for a Week 4 and Month 3 follow-up visit. At the Month 3 follow-up visit, if patients are not showing stability or improvement, they may be offered either thermal laser or Photodynamic Therapy. They will remain in the study and remain eligible for a repeat injection of Anecortave Acetate at the Month 6 visit.

Patients will then been seen at Month 6 for a Re-treatment Evaluation Visit. If their condition is stable, they will be offered re-injection with the same study medication they received earlier. If Patients are not showing stability or improvement at the Month 6 visit, they may be offered thermal laser or Photodynamic Therapy in conjunction with the Anecortave Acetate injection.

If the patient is re-injected at the 6 month visit, the schedule of follow-up visits will repeat as before for the next 18 months. If the patient opts out of the re-injection, they will be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of rubeosis iridis in patients with retinal ischemia.
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 Study Eye on the ETDRS visual acuity chart.
4. Visual acuity of 20/800 or better Fellow Eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within last 2 months.
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document CNV (including difficulty with venous access.
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study.
9. Patient has had insertion of scleral buckle in the study eye.
10. Patient has received radiation treatment.
11. Patient is pregnant or nursing.
12. Patient is on intravenous or subcutaneous anticoagulant therapy, or is on oral anticoagulant therapy (with the exception of aspirin and antiplatelet therapy) and cannot take a 5-day interruption in therapy prior to each depot or sham administration.
13. Patient has evidence of scleral thinning seen at the time of external eye exam or at the time of depot or sham administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
tyo investigate the use of anecortave acetate in rubeosis iridis | 24 months

SECONDARY OUTCOMES:
mean change in VA(ETDRS) from baseline to 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States